CLINICAL TRIAL: NCT02565498
Title: Phase III Study of Preoperative vs Postoperative Intensity Modulated Radiation Therapy For Truncal/Extremity Soft Tissue Sarcoma
Brief Title: Preoperative vs Postoperative IMRT for Extremity/Truncal STS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCREB # 15-070
Record Dates: First submitted 2015-09-18; First posted 2015-10-01 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Adult Soft Tissue Sarcoma
Keywords: Soft tissue sarcoma; Extremity; Preoperative radiotherapy; Postoperative radiotherapy
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preoperative Radiation Therapy (Arm A) (Other): Preoperative intensity modulated radiation therapy followed by surgery
  Interventions: Radiation: Preoperative intensity modulated radiation therapy
- Postoperative Radiation Therapy (Arm B) (Experimental): Surgery followed by postoperative intensity modulated radiation therapy
  Interventions: Radiation: Postoperative intensity modulated radiation therapy

INTERVENTIONS:
Radiation: Preoperative intensity modulated radiation therapy — 50 Gy delivered in 25 fractions 4-6 weeks prior to surgical excision
  Arms: Preoperative Radiation Therapy (Arm A)
Radiation: Postoperative intensity modulated radiation therapy — Surgery followed by 50 Gy delivered in 25 fractions within 6 weeks of surgery for patients with negative margins; for patients with positive margins a boost of 16 Gy in 8 fractions will be added.
  Arms: Postoperative Radiation Therapy (Arm B)

SUMMARY:
This study is designed to determine if preoperative image guided radiation therapy (IGRT) delivered using intensity modulated radiation therapy (IMRT) followed by surgery results in similar short-term wound healing complications as surgery followed by postoperative IGRT in patients with extremity or truncal soft tissue sarcoma. Half of the patients will receive preoperative radiotherapy, half will receive postoperative radiotherapy.

DETAILED DESCRIPTION:
Perioperative RT in addition to surgery is widely accepted as standard management for soft tissue sarcoma (STS) of the extremity and trunk. However, controversy remains as to whether RT should be delivered preoperatively or postoperatively. While both confer similar rates of local control, preoperative RT leads to a decrease in late tissue morbidities such as fibrosis, limb edema, joint stiffness and fracture as compared to postoperative RT. The reasons for this are likely multifactorial, but are in part related to total dose delivered (50 Gray (GY) preoperatively and 60-66 Gy postoperatively) and, based on a previous National Cancer Institute (Canada) Phase III randomized controlled trial, the much larger volume treated in the postoperative setting compared to that in the preoperative setting. The optimal radiation dose used in the postoperative setting is unknown but has been developed empirically and doses of 60-66 Gy are generally employed.However, investigators in Norway/Sweden and France have found equivalent local control rates for patients with negative surgical margins treated with 50 GY postoperativelyThe main concern with preoperative RT has centered on the risk of an increased rate of delayed wound healing and major wound complications. Although some studies suggest it may be possible to reduce the incidence of acute wound healing complications associated with pre-operative radiation than previously seen in the 2D RT era, this has yet to be tested in the phase III setting. IG-IMRT allows a much higher degree of conformality and accurate delivery of dose to the tumour while sparing surrounding normal tissue. This may allow similar rates of acute wound healing complications for pre- and postoperative RT in the treatment of STS.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven soft tissue sarcoma of the extremity or trunk following review by local reference pathologist.
2. Deemed appropriate for preoperative or postoperative radiotherapy and conservative surgery following patient assessment by a radiation oncologist and surgical oncologist.
3. Lesion is primary or locally recurrent. Patient may have undergone excisional biopsy with positive margins at a referring hospital and are eligible following discussion among the surgical oncologists and radiation oncologists that IMRT is an acceptable treatment for that case.
4. Eastern Cooperative Oncology Group (ECOG) score 0-3
5. Patient is aged 18years or older.
6. Patient is able to provide informed consent
7. Patient is available for treatment and follow-up.

Exclusion Criteria:

1. Benign histology.
2. Prior malignancy within the previous five years or concurrent malignancy with the exception of adequately treated basal cell carcinoma of the skin or carcinoma in-situ of the cervix.
3. Prior radiotherapy to the target site
4. Planned chemotherapy for (neo)adjuvant treatment
5. Conservative surgery to the target site
6. Presence of regional nodal disease or unequivocal distant metastases.
7. Other major medical illness deemed to preclude safe administration of protocol treatment or required follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute wound healing complications | 120 days post surgery
  * Secondary operations required for wound treatment (debridement, secondary closure procedures such as rotationplasty, free flaps or skin grafts);
  * Readmission to hospital for wound care;
  * Invasive procedures required for wound care (drainage of hematoma, seroma or infected wound collection);
  * Deep wound packing required at any time (deep packing defined as packing deep to dermis in an area of dehisced wound) to an area of the wound measuring at least 2 cm in length;
  * Prolonged dressing changes, including packing of the wound for greater than six weeks from wound breakdown;
  * Repeat surgery for revision of a split thickness skin graft or requirement for wet dressings for longer than four weeks. (It is permissible for a patient to protect a totally epithelialized skin graft with a dry dressing without declaring a major wound complication)
  * Use of vacuum-assisted closure (VAC)

SECONDARY OUTCOMES:
Acute Radiation Toxicity | Once per week from the start of radiotherapy until its completion (5 weeks in total), then 1 week preop for Group 1; 4 weeks post completion of treatment for Group 2
  Acute radiation skin toxicity will be documented according to the Radiotherapy Oncology Group (RTOG) Acute Radiation Morbidity Scoring Criteria.
Late Radiation Toxicity- RTOG Late Radiation Morbidity | Every 3 months, from 3 months postop for Group 1 and 3 months post RT for Group 2, for 2 years, then 4 monthly for 1 year, then 6 monthly to 5 years.
  Late radiation morbidity to skin, subcutaneous tissue, bone and joints will be documented according to the RTOG/EORTC Late Radiation Morbidity Scoring Scheme.
Late Radiation Toxicity- Common Toxicity Criteria | Every 3 months, from 3 months postop for Group 1 and 3 months post RT for Group 2, for 2 years, then 4 monthly for 1 year, then 6 monthly to 5 years.
  Late radiation morbidity to skin, subcutaneous tissue, bone and joints will be documented according to the Common Toxicity Criteria v4.0
Late Radiation Toxicity- Limb Edema | Every 3 months, from 3 months postop for Group 1 and 3 months post RT for Group 2, for 2 years, then 4 monthly for 1 year, then 6 monthly to 5 years.
  Peripheral limb edema will be documented according to the Late Limb Edema Scoring Criteria.
Limb Function | Within 14 days of randomization, then at 3 and 6 months, 1, 2, 3 and 5 years postop.
  Limb function will be documented according to the Musculoskeletal Tumor Society Rating Scale.
Patient function | Within 14 days of randomization, then at 3 and 6 months, 1, 2, 3 and 5 years postop.
  Patient function will be documented according to the patient completed Toronto Extremity Salvage Score (TESS)
Overall Survival | Surgery Date until 5 years postoperative or death, whichever occurs first
  Overall patient survival in months during the study period
Local recurrence-free survival | Surgery date until 5 years postoperative or local recurrence, whichever occurs first.
  Patient survival without a local recurrence in months during the study period.
Metastasis-free survival | Surgery date until 5 years postoperative or systemic recurrence, whichever occurs first.
  Patient survival without systemic metastases in months during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ferguson, MD, FRCSC, Principal Investigator — MOUNT SINAI HOSPITAL; Peter Chung, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (8):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Canada (4):
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No